CLINICAL TRIAL: NCT03861910
Title: Dietary Choice for the Management of Cow's Milk Allergy Influences the Acquisition of Oral Tolerance and the Occurrence of Other Allergic Manifestations
Brief Title: Dietary Choice for the Management of Cow's Milk Allergy Influences Other Allergic Manifestations
Acronym: ATMAII
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Associate Professor, Federico II University
Other Study IDs: 109n19
Record Dates: First submitted 2019-02-21; First posted 2019-03-04 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Allergy Milk; Allergy;Food; Allergic Asthma; Allergic Conjunctivitis; Allergy Skin
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity; Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- extensively hydrolyzed casein formula+LGG: subjects with IgE mediated cow milk allergy treated with extensively hydrolyzed casein formula plus Lactobacillus rhamnosus GG as exclusion diet
  Interventions: Dietary Supplement: hypoallergenic formulas
- extensively hydrolyzed whey formula;: subjects with IgE mediated cow milk allergy treated with extensively hydrolyzed whey formula as exclusion diet
  Interventions: Dietary Supplement: hypoallergenic formulas
- hydrolyzed rice formula: subjects with IgE mediated cow milk allergy treated with hydrolyzed rice formula as exclusion diet
  Interventions: Dietary Supplement: hypoallergenic formulas
- soy based formula: subjects with IgE mediated cow milk allergy treated with soy based formula as exclusion diet
  Interventions: Dietary Supplement: hypoallergenic formulas
- amino-acid based formula: subjects with IgE mediated cow milk allergy treated with amino-acid based formula as exclusion diet
  Interventions: Dietary Supplement: hypoallergenic formulas

INTERVENTIONS:
Dietary Supplement: hypoallergenic formulas — hypoallergenic formulas used for cow milk allergy treatment

SUMMARY:
Food allergy is a common chronic condition in childhood. Recent studies have suggested that the natural history of food allergy has changed during the last two decades, with an increased prevalence, severity of clinical manifestations, and risk of persistence into later ages. The increased food allergy prevalence in children has an important economic impact, with significant direct costs for the healthcare system and even larger costs for the families of food-allergic patients. In addition, children with food allergies are at increased risk to develop other allergic manifestations later in life. According to a recent study, children with a food allergy are 2 to 4 times more likely to develop other atopic manifestations such as asthma (4.0 times), atopic eczema (2.4 times), and respiratory allergies (3.6 times), compared to children without a food allergy. Cow's milk allergy is among the most common food allergy in early childhood, with an estimated prevalence of 2% to 3%. It has been previously showed that in children with cow milk allergy, an extensively hydrolysed casein formula supplemented with the probiotic Lactobacillus rhamnosus GG induced higher tolerance rates compared to extensively hydrolysed casein formula without Lactobacillus rhamnosus GG and other formulas. These findings were consistent with those of a 1-year follow-up study performed in the US that showed better outcomes using an extensively hydrolysed casein formula+Lactobacillus rhamnosus GG vs. an extensively hydrolysed casein formula or amino acid-based formula for the first-line dietary management of cow milk allergy. In addition it has been recently demonstrated that extensively hydrolysed casein formula + Lactobacillus rhamnosus GG reduces the incidence of other atopic manifestations and hastens the development of oral tolerance in children with IgE-mediated cow milk allergy.

The present randomized controlled trial (RCT) was designed to test whether different dietary interventions could influence the occurrence of other atopic manifestations in children with IgE-mediated cow milk allergy.

ELIGIBILITY:
Inclusion Criteria:

* age 1-12 months
* IgE-mediated CMA

Exclusion Criteria:

* cow's milk protein-induced anaphylaxis,
* food protein induced enterocolitis syndrome,
* other food allergies,
* other allergic diseases,
* non-CMA-related atopic eczema,
* eosinophilic disorders of the gastrointestinal tract,
* chronic systemic diseases,
* congenital cardiac defects,
* active tuberculosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* chronic pulmonary diseases,
* malformations of the gastrointestinal and/or respiratory tract,
* administration of prebiotics or probiotics during the 4 weeks before enrolment.

Ages: 1 Month to 12 Months | Sex: All
Age Groups: Child
Study Population: Children who were consecutively observed at a FP office because the recent occurrence of signs and symptoms possibly related to IgE-mediated CMA were sent to our tertiary centre for paediatric allergy for possible inclusion in the study. Only subjects who met the inclusion criteria will be invited to participate to the study.Written informed consent will be obtained from the parents of each subject. Anamnestic, demographic, anthropometric and clinical data, as well as information on socio-demographic factors, family and living conditions, parental history of allergic diseases, maternal smoking during pregnancy, environmental tobacco smoke exposure, number of siblings, and pet ownership were obtained from the parents and recorded in a clinical database. For children with sure diagnosis of IgE-mediated CMA during a 3-year follow-up,3 visits every 12 months will be performed. Stool samples for metagenomics and metabolomics and blood sample for epigenetics studies will be collected.
Sampling Method: Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Rate of subjects with occurrence of other of allergic manifestations | 3 years
  To evaluate the effect of different dietary strategies on the occurrence of eczema, urticaria, asthma and rhinoconjunctivitis in children with IgE-mediated cow milk allergy

SECONDARY OUTCOMES:
Rate of subjects with tolerance acquisition to cow's milk | 3 years
  To evaluate the tolerance acquisition to cow's milk
Change in metagenomics and metabolomics | 3 years
  16S rRNA gene amplicon sequencing
Epigenetic modifications in cytokines genes | 3 years
  Serum levels (pg/ml) of interleukin 4, interleukin 5, interleukin 10, interferon gamma, FOXP3 in children with cow's milk allergy
Epigenetic modifications in cytokines genes | 3 years
  Methylation rate (%) of interleukin 4, interleukin 5, interleukin 10, interferon gamma, FOXP3 in children with cow's milk allergyFOXP3 in children with cow's milk allergy
Rate of subjects with occurrence of other of allergic manifestations | after 4 to 6 years follow-up
  To evaluate the effect of different dietary strategies on the occurrence of eczema, urticaria, asthma and rhinoconjunctivitis in children with IgE-mediated cow milk allergy
Rate of subjects with tolerance acquisition to cow's milk | after 4 to 6 years follow-up
  To evaluate the tolerance acquisition to cow's milk
Rate of subjects with any autoimmune disease | 6 years
  To evaluate the occurrence of type 1 diabetes, celiac disease, juvenile idiopathic arthritis, thyroiditis, inflammatory bowel diseases

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided